CLINICAL TRIAL: NCT02305355
Title: Efficacy and Safety of Prescription Omega-3 Fatty Acid Added to Stable Statin Therapy in Patients With Type 2 Diabetes and Hypertriglyceridemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kuhnil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-OM-9412
Record Dates: First submitted 2014-11-25; First posted 2014-12-02 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes Mellitus, Type 2; Hypertriglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pravastatin; Simvastatin; Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3-acids ethylesters 90 4g, any statin (Experimental)
  Interventions: Drug: Omega-3-acids ethylesters 90 4g; Drug: Pravastatin, Simvastatin, Atorvastatin, Rosuvastatin
- any statin (Active Comparator)
  Interventions: Drug: Pravastatin, Simvastatin, Atorvastatin, Rosuvastatin

INTERVENTIONS:
Drug: Omega-3-acids ethylesters 90 4g
  Other Names: Omacor Soft Capsule 4g
  Arms: Omega-3-acids ethylesters 90 4g, any statin
Drug: Pravastatin, Simvastatin, Atorvastatin, Rosuvastatin

SUMMARY:
Assess efficacy and safety of Omacor® 4g with statin treatment for lowering TG levels in subjects with type 2 Diabetes combined with hyperlipidemia

ELIGIBILITY:
Inclusion Criteria:

* LDL-C < 100mg/dL, TG > 150mg/dL, patients on statin treatment for at least 6 weeks prior to randomization.
* Type 2 Diabetes
* HbA1c ≤ 10.0

Exclusion Criteria:

* Type 1 Diabetes
* Patients with PPAR gamma agonist therapy
* Patients with acute MI, Unstable angina within 6 months
* History of malignant tumor within 2 years
* Women with pregnant, breast-feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The mean percent change of Triglyceride(TG) | from baseline at week 16

SECONDARY OUTCOMES:
The mean percent change of Total Cholesterol(TC) | from baseline at week 16
The mean percent change of LDL-C | from baseline at week 16
The mean percent change of HDL-C | from baseline at week 16
The mean percent change of HBA1c | from baseline at week 16
The mean percent change of FPG | from baseline at week 16
The mean percent change of hs-CRP | from baseline at week 16
The mean percent change of PAI-1 | from baseline at week 16
The mean percent change of Apolipoprotein A1 | from baseline at week 16
The mean percent change of apolipoprotein B | from baseline at week 16

CONTACTS AND LOCATIONS:
Locations (1):
- Bucheon St. Mary's Hospital, Bucheon-si, South Korea

REFERENCES:
- [Derived] Son JW, Kim CH, Nam MS, Park IB, Yoo SJ. Efficacy and Safety of Prescription Omega-3 Fatty Acids Added to Stable Statin Therapy in Korean Patients with Type 2 Diabetes and Hypertriglyceridemia: a Randomized Controlled Trial. J Lipid Atheroscler. 2019 Sep;8(2):221-231. doi: 10.12997/jla.2019.8.2.221. Epub 2019 Jul 4. PMID 32821712